CLINICAL TRIAL: NCT06815393
Title: Comparison of the Analgesic Effect of Intrathecal Morphine and Bilateral Transversus Abdominis Plane Block in Patients Undergoing Elective Abdominal Hysterectomy
Brief Title: COMPARISON of the EFFECT of TWO DIFFERENT ANALGESIS TECHNIQUES in ABDOMINAL HYSTERECTOMY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emirhan Akarsu, Resaerch Resident, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2024-04/07
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Hysterectomy
Keywords: abdominal hysterectomy; intratechal morphine; transversalis fascia plane block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Intratechal Morphine (Active Comparator)
  Interventions: Other: Intratechal Morphine
- Group Transversalis Fascia Plane Block (Active Comparator)
  Interventions: Other: Transversalis Fascia Plane Block

INTERVENTIONS:
Other: Intratechal Morphine — Prior to induction, the patient will be positioned seated, and morphine will be slowly injected intrathecally at a dose of 5 μg/kg, adjusted to the L4-L5 or L3-L4 intervertebral space using a 27G pencil point spinal needle. The injection will be administered over approximately 10 seconds
  Arms: Group Intratechal Morphine
Other: Transversalis Fascia Plane Block — Prior to induction, patients will be positioned supine, and bilateral transversus abdominis plane (TAP) block will be performed with the aid of ultrasound. As the blocking agent, 20 cc of 0.25% bupivacaine will be used bilaterally.
  Arms: Group Transversalis Fascia Plane Block

SUMMARY:
Hysterectomy is one of the most commonly performed surgical procedures after cesarean section in many countries worldwide, especially among women of reproductive age. Postoperative pain is typically managed with oral and parenteral narcotics. Patient-controlled analgesia (PCA) is an effective pain management method that provides advantages such as faster pain relief, better dosage control, and elimination of the need for timer adjustments. Facilitating the recovery process and optimizing postoperative pain management are crucial components of perioperative care. To minimize systemic opioid requirements and opioid-related side effects, multimodal analgesia combining local anesthesia, peripheral, and non-opioid analgesics has become increasingly popular.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 65 years classified as ASA 1 and ASA 2.

Exclusion Criteria:

* Patients with allergies to the active substance, those with severe liver or renal insufficiency, a history of long-term nonsteroidal anti-inflammatory drug (NSAID) and opioid analgesic use, a history of gastrointestinal bleeding, peptic ulcer or inflammatory bowel disease, a history of diabetes or other neuropathic conditions, preoperative atrioventricular block and bradycardia, underlying serious respiratory diseases, a history of psychiatric disorders, patients classified as ASA stage 3 or higher, patients weighing less than 40 kg, patients unable to use the patient-controlled analgesia (PCA) device, and patients who need to discontinue the study medication during surgery for any reason will be excluded from the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperatve Opioid Consumption | postoperatively 24 hours
  The primary aim of this study is to compare the analgesic efficacy of intrathecal morphine and bilateral transversalis fascia plane block in patients undergoing elective abdominal hysterectomy, in terms of morphine consumption during the first 24 hours postoperatively

SECONDARY OUTCOMES:
Postoperative Pain Scores at movement and rest | postoperatively 24 hours
  evaluation of pain scores during movement and rest within 24 hours postoperatively using Visual Analogue Scale
Quality of recovery 24 hours after the surgery assessed using QoR-40 questionnaire | postoperative 24 hour
  Evaluation of quality of recovery 24 hours after the surgery assessed using QoR-40 questionnaire
Advers Event | postoperative 24 hour
  incidence of side effects (nause, vomiting, urinary retention) for 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)